CLINICAL TRIAL: NCT05435612
Title: Evaluation of Rehabilitation Results in the Single-sided Deafness/Asymmetrical Hearing Loss With Cochlear Implantation
Brief Title: Evaluation of Rehabilitation Results in the Single-sided Deafness With Cochlear Implantation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, YangShiming, College of Otolaryngology Head and Neck Surgery, Chinese PLA General Hospital, Chinese PLA General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SSD-2022-01
Record Dates: First submitted 2022-06-06; First posted 2022-06-28 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Unilateral Deafness
MeSH Terms: conditions — Hearing Loss, Unilateral | interventions — Cochlear Implants

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- single-sided deafness group（SSD Group） (Experimental): The single-sided group（SSD group）consists of 20 SSD patients voluntarily enrolled in the study and plan to undergo cochlear implantation.
  Interventions: Device: cochlear implant
- asymmetric hearing loss group（AHL Group） (Experimental): The asymmetric hearing loss group（AHL group）consists of 10 AHL patients voluntarily enrolled in the study and plan to undergo cochlear implantation.
  Interventions: Device: cochlear implant

INTERVENTIONS:
Device: cochlear implant — Patients enrolled in the study undergo the cochlear implant surgery.

SUMMARY:
Single-sided deafness (SSD) refers to severe to profound sensorineural hearing loss on one side (average pure-tone hearing threshold≥70 dB HL at 0.5, 1, 2, and 4kHz) while the opposite side maintains normal hearing or mild hearing loss (30 dB HL). Asymmetrical hearing loss (AHL) refers to severe to profound sensorineural hearing loss in the bad ear (average pure-tone hearing threshold≥70 dB HL at 0.5, 1, 2, and 4kHz) and mild to moderate hearing loss in the contralateral ear. Moderate hearing loss (30≤mean pure-tone hearing threshold≤55dBHL). It is generally acknowledged that SSD is a particular clinical manifestation of AHL. The number of people who have hearing loss accounts for 5.3% of the total population, with children for 9%. According to the Second National Sampling Survey on Disabled Persons, China has 27.8 million people with hearing disabilities. The incidence of SSD adults in the United States is 7.2%, with 60,000 new cases per year, compared with 7,500 new patients with SSD annually in the UK. The incidence of SSD in neonates is 0.04%-0.34%, and it ranges from 0.1% to 0.5% in children and adolescents. The etiology of congenital SSD is primarily unknown, which is related to genes. Among the causes of acquired SSD, sudden deafness is the most common. Other causes include head trauma, Meniere's disease, labyrinthitis, unilateral acoustic neuroma, middle ear surgery, ototoxic drug exposure, Virus infection, noise-induced deafness, senile deafness, etc.

SSD and AHL impede intellectual development and speech development in children and adolescents, which is associated with the side of hearing loss. For example, children with right-sided hearing loss have relatively poor language learning, logical thinking, and divergent thinking. In contrast, children with left-sided hearing loss have weaker analytical, comprehensive and visual memory abilities and relatively poor spatial imagination and visual-motor coordination. In addition, the lack of long-term monaural listening and sound source localization makes SSD children require excessive concentration, which is prone to fatigue and behavioral problems, and their academic performance is lower than that of normal children.

DETAILED DESCRIPTION:
Current options for hearing interventions for patients with SSD are air conduction hearing aids, bone conduction hearing aids and cochlear implants. Attributed to the United States Food and Drug Administration (FDA) approval of one manufacturer's CI for patients aged five years and older with SSD in 2019, CI has been considered by the growing population. However, few studies on CI in patients with SSD, especially in China. Therefore, the study aims to evaluate the efficacy of CI in SSD patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 12 years old and above
2. Language ability: postlingual deafness, able to cooperate with sentence test in noise
3. Normal mental, intelligence and motor development
4. Patients who meet the diagnosis of single-sided deafness and asymmetric hearing loss

Exclusion Criteria:

1. Cochlear malformation (except large vestibular aqueduct syndrome)
2. Retrocochlear lesions
3. Incomplete implantation of cochlear implant electrodes
4. Non-Chinese Mandarin communication

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-07-05 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
speech recognition | The tests are conducted before the cochlear implantation.
  Both speech recognition score and speech recognition threshold are conducted to assess the auditory sensitivity and articulation of the spoken language. That is to evaluate the subjects' ability to recognize and understand speech in actual communication.
speech recognition | The tests are conducted 1 months after CI activation.
  Both speech recognition score and speech recognition threshold are conducted to assess the auditory sensitivity and articulation of the spoken language. That is to evaluate the subjects' ability to recognize and understand speech in actual communication.
speech recognition | The tests are conducted 3 months after CI activation.
  Both speech recognition score and speech recognition threshold are conducted to assess the auditory sensitivity and articulation of the spoken language. That is to evaluate the subjects' ability to recognize and understand speech in actual communication.
speech recognition | The tests are conducted 6 months after CI activation.
  Both speech recognition score and speech recognition threshold are conducted to assess the auditory sensitivity and articulation of the spoken language. That is to evaluate the subjects' ability to recognize and understand speech in actual communication.
speech recognition | The tests are conducted 12 months after CI activation.
  Both speech recognition score and speech recognition threshold are conducted to assess the auditory sensitivity and articulation of the spoken language. That is to evaluate the subjects' ability to recognize and understand speech in actual communication.
sound localization | The test is conducted before the cochlear implantation.
  180° (horizonal) sound localization test is conducted to assess the sound source localization ability (pre-/post-operation).
sound localization | The test is conducted 1 months after CI activation.
  180° (horizonal) sound localization test is conducted to assess the sound source localization ability (pre-/post-operation).
sound localization | The test is conducted 3 months after CI activation.
  180° (horizonal) sound localization test is conducted to assess the sound source localization ability (pre-/post-operation).
sound localization | The test is conducted 6 months after CI activation.
  180° (horizonal) sound localization test is conducted to assess the sound source localization ability (pre-/post-operation).
sound localization | The test is conducted 12 months after CI activation.
  180° (horizonal) sound localization test is conducted to assess the sound source localization ability (pre-/post-operation).
Objective electroencephalography-based assessment(EEG) | The test is conducted before the cochlear implantation.
  EEG is a non-invasive objective assessment technique that records brain activity along with specific neural pathways. we utilize cortical auditory evoked potential (CAEP) and event-related potentials(ERP) to obtain time-domain analysis.
Objective electroencephalography-based assessment(EEG) | The test is conducted 1 months after CI activation.
  EEG is a non-invasive objective assessment technique that records brain activity along with specific neural pathways. we utilize cortical auditory evoked potential (CAEP) and event-related potentials(ERP) to obtain time-domain analysis.
Objective electroencephalography-based assessment(EEG) | The test is conducted 3 months after CI activation.
  EEG is a non-invasive objective assessment technique that records brain activity along with specific neural pathways. we utilize cortical auditory evoked potential (CAEP) and event-related potentials(ERP) to obtain time-domain analysis.
Objective electroencephalography-based assessment(EEG) | The test is conducted 6 months after CI activation.
  EEG is a non-invasive objective assessment technique that records brain activity along with specific neural pathways. we utilize cortical auditory evoked potential (CAEP) and event-related potentials(ERP) to obtain time-domain analysis.
Objective electroencephalography-based assessment(EEG) | The test is conducted 12 months after CI activation.
  EEG is a non-invasive objective assessment technique that records brain activity along with specific neural pathways. we utilize cortical auditory evoked potential (CAEP) and event-related potentials(ERP) to obtain time-domain analysis.

SECONDARY OUTCOMES:
THI (Tinnitus Handicap Inventory) | The test is conducted before the cochlear implantation.
  The tinnitus-related questionnaire has a comprehensive understanding of tinnitus from three aspects(functional scale, emotional scale and catastrophic scale).
THI (Tinnitus Handicap Inventory) | The test is conducted 1 months after CI activation.
  The tinnitus-related questionnaire has a comprehensive understanding of tinnitus from three aspects(functional scale, emotional scale and catastrophic scale).
THI (Tinnitus Handicap Inventory) | The test is conducted 3 months after CI activation.
  The tinnitus-related questionnaire has a comprehensive understanding of tinnitus from three aspects(functional scale, emotional scale and catastrophic scale).
THI (Tinnitus Handicap Inventory) | The test is conducted 6 months after CI activation.
  The tinnitus-related questionnaire has a comprehensive understanding of tinnitus from three aspects(functional scale, emotional scale and catastrophic scale).
THI (Tinnitus Handicap Inventory) | The test is conducted 12 months after CI activation.
  The tinnitus-related questionnaire has a comprehensive understanding of tinnitus from three aspects(functional scale, emotional scale and catastrophic scale).
SSQ12 (Speech, Spatial and Qualities of Hearing Scale) | The test is conducted before the cochlear implantation.
  SSQ12 questionnaire investigate the listening situation in daily environment, which is divided into three dimensions: speech perception, spatial hearing and auditory quality.
SSQ12 (Speech, Spatial and Qualities of Hearing Scale) | The test is conducted 1 months after CI activation.
  SSQ12 questionnaire investigate the listening situation in daily environment, which is divided into three dimensions: speech perception, spatial hearing and auditory quality.
SSQ12 (Speech, Spatial and Qualities of Hearing Scale) | The test is conducted 3 months after CI activation.
  SSQ12 questionnaire investigate the listening situation in daily environment, which is divided into three dimensions: speech perception, spatial hearing and auditory quality.
SSQ12 (Speech, Spatial and Qualities of Hearing Scale) | The test is conducted 6 months after CI activation.
  SSQ12 questionnaire investigate the listening situation in daily environment, which is divided into three dimensions: speech perception, spatial hearing and auditory quality.
SSQ12 (Speech, Spatial and Qualities of Hearing Scale) | The test is conducted 12 months after CI activation.
  SSQ12 questionnaire investigate the listening situation in daily environment, which is divided into three dimensions: speech perception, spatial hearing and auditory quality.
QLBHE (Quality of Life for Bilateral Hearing Effect) | The test is conducted before the cochlear implantation.
  QLBHE questionnaire is to evaluate the effect of bilateral listening in daily life after the use of assisted hearing devices.
QLBHE (Quality of Life for Bilateral Hearing Effect) | The test is conducted 1 months after CI activation.
  QLBHE questionnaire is to evaluate the effect of bilateral listening in daily life after the use of assisted hearing devices.
QLBHE (Quality of Life for Bilateral Hearing Effect) | The test is conducted 3 months after CI activation.
  QLBHE questionnaire is to evaluate the effect of bilateral listening in daily life after the use of assisted hearing devices.
QLBHE (Quality of Life for Bilateral Hearing Effect) | The test is conducted 6 months after CI activation.
  QLBHE questionnaire is to evaluate the effect of bilateral listening in daily life after the use of assisted hearing devices.
QLBHE (Quality of Life for Bilateral Hearing Effect) | The test is conducted 12 months after CI activation.
  QLBHE questionnaire is to evaluate the effect of bilateral listening in daily life after the use of assisted hearing devices.
NCIQ (Nijmegen Cochlear Implant Questionnaire) | The test is conducted before the cochlear implantation.
  The questionnaire evaluates the quality of life of patients from three dimensions: physiological function, psychological function and social function.
NCIQ (Nijmegen Cochlear Implant Questionnaire) | The test is conducted 1 months after CI activation.
  The questionnaire evaluates the quality of life of patients from three dimensions: physiological function, psychological function and social function.
NCIQ (Nijmegen Cochlear Implant Questionnaire) | The test is conducted 3 months after CI activation.
  The questionnaire evaluates the quality of life of patients from three dimensions: physiological function, psychological function and social function.
NCIQ (Nijmegen Cochlear Implant Questionnaire) | The test is conducted 6 months after CI activation.
  The questionnaire evaluates the quality of life of patients from three dimensions: physiological function, psychological function and social function.
NCIQ (Nijmegen Cochlear Implant Questionnaire) | The test is conducted 12 months after CI activation.
  The questionnaire evaluates the quality of life of patients from three dimensions: physiological function, psychological function and social function.

CONTACTS AND LOCATIONS:
Overall Officials: Shiming Yang, MD, Study Director — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China